CLINICAL TRIAL: NCT01775319
Title: Evaluation of Human Zinc Absorption From Wheat-based Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: HarvestPlus (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HNL/CTC_Zn_wheat; KEK-ZH-2012-0483 (Other: KEK-Zurich)
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Zinc Deficiency
Keywords: Zinc

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biofortified wheat (Active Comparator): Biofortified wheat
  Interventions: Dietary Supplement: Biofortified wheat
- Control wheat (Placebo Comparator): Control wheat with low level of Zn
  Interventions: Dietary Supplement: Placebo
- Fortified wheat (Active Comparator): Wheat fortified before consumption
  Interventions: Dietary Supplement: Fortified wheat

INTERVENTIONS:
Dietary Supplement: Biofortified wheat — Extrinsic label 67Zn (ZnSO4) 0.2mg 70Zn added to the IV dose
  Other Names: Esperia
  Arms: Biofortified wheat
Dietary Supplement: Fortified wheat — Extrinsic label 67Zn (ZnSO4) 0.2mg 70Zn added to the IV dose
  Arms: Fortified wheat
Dietary Supplement: Placebo
  Arms: Control wheat

SUMMARY:
Study part 1 and 2 Assessment of Zn absorption from regular and biofortified wheat: stable isotope absorption studies in women of childbearing age consuming test meals prepared from either the biofortified Zn wheat, regular wheat or post-harvest fortified wheat at two different extraction rates.

Study part 3 Assessment of Zn absorption from intrinsically and extrinsically labeled wheat: stable isotope absorption studies in women of childbearing age, or men, consuming test meals prepared from either intrinsically labeled Zn biofortified wheat, regular wheat or post-harvest fortified wheat extrinsically labeled immediately before consumption.

DETAILED DESCRIPTION:
The overall goal of study part 1 and 2 is to evaluate and compare the fractional and absolute Zn absorption from biofortified wheat cultivar (60 ppm Zn) to regular wheat (28 ppm Zn) and to post harvest fortified wheat (60 ppm Zn) for a total of 3 test meals per study. The studies will be conducted with products based on wheat with high extraction rate (study part 1) and medium extraction rate (study part 2) in two separate groups of women of childbearing age.

The goal of study part 3 is to investigate the difference of absorption measurements between intrinsically and extrinsically labeled biofortified wheat. The label of the test meals will have the same nature as the fortificant itself (extrinsic vs intrinsic), for a total of 3 test meals.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old (Study part 1 and 2). Female or male, 18 to 45 years old (Study part 3)
* Body Mass Index in the range of 18.5 to 25 kg/m2
* Signed informed consent

Exclusion Criteria:

* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, anemia, hepatitis, hypertension, cancer or cardiovascular diseases (according to the subjects own statement)
* Gluten intolerance, celiac disease
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Vegans
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st test meal administration
* Smoking
* Pregnancy (Urine pregnancy test shall be performed before each test meal administration)
* Lactating
* Earlier participation in a study using Zn stable isotopes or participation in any other clinical study within the last 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Fractional zinc absorption from different wheat-based test meals | 3 months
  Fractional zinc absorption (in %) will be assessed with stable isotopes of zinc using a double isotope technique.

SECONDARY OUTCOMES:
Zn and C-reactive protein concentration in plasma | 3 months

OTHER OUTCOMES:
Creatinin | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — Swiss Federal Institute of Technology

REFERENCES:
- [Derived] Signorell C, Zimmermann MB, Cakmak I, Wegmuller R, Zeder C, Hurrell R, Aciksoz SB, Boy E, Tay F, Frossard E, Moretti D. Zinc Absorption From Agronomically Biofortified Wheat Is Similar to Post-Harvest Fortified Wheat and Is a Substantial Source of Bioavailable Zinc in Humans. J Nutr. 2019 May 1;149(5):840-846. doi: 10.1093/jn/nxy328. PMID 31004128